CLINICAL TRIAL: NCT06984536
Title: Reduced-dose Anti-thymocyte Globulin Plus Mini-dose Post-transplant Cyclophosphamide for GVHD Prevention in Haploidentical Donor HCT for Hematologic Malignancy
Brief Title: Reduced ATG Plus Mini PTCy for GVHD Prophylaxis in Haplo-SCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Peking University People's Hospital, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Lower ATG plus miniPTCy
Record Dates: First submitted 2025-05-03; First posted 2025-05-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndrome; Acute Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reduced ATG puls mini PTCy (Experimental): Patients recieved ATG 7.5mg/kg plus PTCy 14.5mg/kg on day +3 and +4 for GVHD prophylaxis in haplo-SCT
  Interventions: Drug: Reduced ATG plus mini PTCy

INTERVENTIONS:
Drug: Reduced ATG plus mini PTCy — The conditioning protocol comprises cytarabine (Ara-C) (4 g/m2/day, days -9), busulfan (Bu) (3.2 mg/kg/day, days -8 to -6), cyclophosphamide (Cy) (1.8 g/m2/kg, days -5 and -4), simustine (250 mg/m2, day -3) and r-ATG (total 7.5mg/kg ,from days -5 to -2). Mini PTCy 14.5mg/kg/day will be given on day +3 and +4.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is regarded as a curative therapy for a variety of hematological malignancies and nonmalignant diseases. However, donor limitations have restricted the widespread use of allo-HSCT for a long period. The development and success of haploidentical allografts worldwide makes "everyone has a donor" a reality. In the past two decades, researchers have established several haploidentical HSCT (haplo-HSCT) protocols based on different approaches to induce immune tolerance. The representative approaches for haplo-HSCT without in vitro. T cell depletion include granulocyte colony-stimulating factor (G-CSF) plus Anti-human Thymocyte Immunoglobulin (ATG) based (Beijing Protocol) and post-transplantation cyclophosphamide based (PT-Cy, Baltimore Protocol) protocols. Both of two protocols have common problems that need to be solved, including infection transplantation related mortality and disease relapse. The main aim of this study is to explore whether the combined protocol can improve the efficacy of haploidentical transplantation further.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AL - CR and/or myelodysplastic syndromes undergoing allogeneic hematopoietic stem cell transplantation for the first time;
2. No gender limit, aged 12 - 65 years;
3. Planned haploidentical donor transplantation, excluding transplantation from maternal and collateral donors;
4. Eastern Cooperative Oncology Group (ECOG) performance status score≤3 points;
5. Baseline organ function tests meet the following criteria:

(1) Left ventricular ejection fraction (LVEF) > 55%; (2) Serum creatinine ≤ 1.5 × upper limit of normal (ULN).

Exclusion Criteria:

1. Patients with severe dysfunction of brain, heart, kidney or liver;
2. Those in refractory malignant status;
3. Patients with other malignancies requiring treatment;
4. Presence of uncontrolled severe active infection clinically;
5. Expected survival period of less than 3 months;
6. History of severe allergic reactions;
7. Pregnant or breastfeeding women; (8)Presence of any condition deemed by the investigator as unsuitable for study enrollment.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Non-relapse mortality | 100 days
  None-relapse mortality within 100 days post transplantation

SECONDARY OUTCOMES:
Regimen related toxicity | 30 days post transplantation
  Regimen related toxicity will be evaluated by Bearman Criteria from the begining of conditioning to 1 month post HSCT. The organ functions that need to be assessed include the heart, liver, kidneys, cystitis, oral mucositis, and the gastrointestinal tract.
Engraftment | Within 30 days post transplant. Myeloid engraftment was deﬁned as the ﬁrst of three consecutive days with an ANC 0.5×109 /L, and platelet engraftment was deﬁned as the day the platelet count met or exceeded 20×10^9 /L without transfusion for a week.
  Myeloid and platelet engraftment
Disease relapse | 1 year post transplantation
  The incidence of disease relapse
Disease free survival | 1 year post transplantation
  The time from the start of transplantation until a patient experiences leukemia relapse or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People'S Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No